CLINICAL TRIAL: NCT05732974
Title: A Machine Learning Approach to Identify Patients With Resected Non-small-cell Lung Cancer With High Risk of Relapse
Acronym: MIRACLE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0519
Record Dates: First submitted 2022-11-14; First posted 2023-02-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer Stage IIIA
Keywords: Machine-learning; Resected early stage Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biomarkers detected on plasma and tissue samples for analysis of circulating and extracellular vesicles-derived microRNAs as well as of free circulating DNA performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resected early stage non small cell lung cancer: Early stage (IA-IIIA) resectable non small cell lung cancer patients receiving surgery
  Interventions: Other: Resected non small cell lung cancer

INTERVENTIONS:
Other: Resected non small cell lung cancer — plasma sample, tissue sample and computed tomography scan images

SUMMARY:
Early-stage non small cell lung cancer represents 20-30% of all non small cell lung cancer and is characterized by a high survival probability after surgical resection. However, considering stage IA-IIIA non small cell lung cancer, a relapse rate of about 50% is observed, with a different survival probability on the basis of tumor node metastasis status, although patients within the same tumor node metastasis stage exhibit wide variations in recurrence rate. There are currently no validated prognostic biomarkers able to identify patients with a high risk of relapse.

DETAILED DESCRIPTION:
This study will use data from an already available cohort of patients enrolled in the Resting study (a project funded by TRANSCAN in 2018) as a training set and data from a new concurrent cohort as validation set.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an early stage of non small cell lung cancer
* Indication of surgical resection
* Patient able to understand and give his consent
* Patient affiliated to the health insurance

Exclusion Criteria:

* Patient with another cancer in the last 5 years
* Patient with an allergy to the contrast medium
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an early stage of non small cell lung cancer with an indication of surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Algorithm for disease free survival | 18 months
  Analysis on a training cohort of resected early-stage non small cell lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Julien MAZIERES, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Julien MAZIERES, Toulouse, France

IPD SHARING:
Plan to Share IPD: No